CLINICAL TRIAL: NCT02938819
Title: Effects of a Goal-oriented Upper-limb Intervention in Patients With Parkinson's Disease
Brief Title: Goal-oriented Intervention in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0062UG
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson's Disease
Keywords: upper limbs; physiotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group received a Goal-oriented upper limb intervention.
  Interventions: Other: Goal-oriented upper-limb intervention
- Control group (Active Comparator): Patients in the control group received a standard upper limb intervention
  Interventions: Other: Standard upper limb intervention

INTERVENTIONS:
Other: Goal-oriented upper-limb intervention — The Goal-oriented upper-limb intervention evaluated patients' expectations and the environmental factors influencing the performance of the specific task were identified for each of the three tasks. Patients were asked to perform the activity at home. After this, the observable target behavior corresponding to the target activity was determined. Then, an occupational and a physical therapist worked together with the patient to identify the assistance required to perform this activity such as human assistance, technical aids, assistive devices or verbal guidance.
  Arms: Experimental group
Other: Standard upper limb intervention — The standard upper limb intervention involved active upper limb range of motion, manual dexterity involving grasp and manipulation of small pieces such as marbles and stretching upper limb exercises.
  Arms: Control group

SUMMARY:
Upper-limb disorders in patients with Parkinson's disease include decreased speed and amplitude of movements, difficulty in sequential tasks, and disrupted execution of fine manipulative hand activities.The aim of the study was to evaluate the effects of home-based goal-oriented upper limb intervention in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative neurological disorders involving progressive impairment in motor, mood and cognitive functions. Movement disorders have a negative impact on individual's ability to perform well-learned motor skills. These include akinesia, bradykinesia, rigidity and tremor at rest.

A goal-planning process should be useful to ensure that patients agree on the goals of rehabilitation. Thus, the purpose of the study was to evaluate the effects of home-based goal-oriented upper limb intervention in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's Disease.
* Stage II-III of disease progression as defined by the Hoehn and Yahr scale.
* Upper limbs impairment

Exclusion Criteria:

* Clinical signs of dementia or psychiatric disturbance.
* Comprehension deficits that prevented them from following verbal commands.
* Visual or acoustic limitations.
* A neurologic condition other than Parkinson's Disease.
* Musculoskeletal disorders and/or if they had previous trauma or fracture of upper extremity.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Goals attainment | Change from baseline goals attainment assessment at 4 weeks.
  Attainment of goals was assessed using the Goal Attainment Scaling, a method for quantifying progress on the achievement of specific goals

SECONDARY OUTCOMES:
Manual dexterity | Change from baseline manual dexterity at 4 weeks
  Manual dexterity was assessed using Purdue Pegboard test (one task with the dominant hand, one with the non-dominant hand, one with both hands and assembly task).
Handgrip strength | Change from baseline handgrip strength at 4 weeks
  Handgrip strength was assessed using a dynamometer
Finger prehension force | Change from baseline finger prehension force at 4 weeks
  Finger prehension force was assessed using a pinch meter

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physical Therapy, Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: Undecided